CLINICAL TRIAL: NCT03266380
Title: Risk Factors and Common Preventive Measures for Ventilator Associated Pneumonia in Patients With Severe Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed mahmoud abdelaziz, specialist at anesthesia and ICU department, Assiut University
Other Study IDs: VAP
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: observational — All patients do an emergency brain computed tomography scan. Intracranial hypertension is treated with mannitol with or without a craniotomy. A third generation cephalosporin (ceftriaxone) and metronidazole are administered as antibiotic prophylaxis for accompanying wound injuries (skin and soft tissue). VAP preventive strategies that are performed in the ICU include daily interruption of sedation and a readiness to extubate assessment, early facilitation of mobility, elevating the head of the bed to 30- 45 degree, change of the ventilator circuit if visibly soiled or malfunctioning, stress ulcer prophylaxis, residual gastric volume monitoring, early parenteral nutrition, and deep venous thrombosis prophylaxis. An infusion of midazolam and propofol is to be used for sedation.

SUMMARY:
The primary objective of this study is to assess the incidence of VAP in patients with TBI and to identify risk factors for developing VAP in this specific patient population (types of co-injuries in patients with multiple trauma or characteristics on admission). The secondary objective is to assess the prevalence of pathogens responsible for early- and late-onset VAP in patients with TBI. The tertiary objective is to discuss the ability of preventive measures to reduce the incidence of VAP

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is a type of nosocomial pneumonia that occurs in patients who receive >48 h of mechanical ventilation (MV). Early onset VAP occurs during the first 4 days of MV and is usually caused by antibiotic-sensitive bacteria. The increased systemic inflammatory response in patients with a head trauma may predispose them to develop early-onset VAP1,2. Late-onset VAP develops 5 days after initiating MV and is caused by multidrug resistant (MDR) pathogens3,4.

Patients with traumatic brain injury (TBI) are at high risk of infection, particularly nosocomial infections, during treatment in the intensive care unit (ICU) 5-7, where the incidence of VAP can be as high as 50%. The duration of MV usually influences the type of organism that causes VAP8. Early-onset VAP is caused by antibiotic-sensitive pathogens, whereas late-onset VAP is caused by MDR bacteria, which are more difficult to treat. The microbiological environment can have a marked influence on VAP isolates, particularly during late-onset VAP, but it also influences early-onset VAP9. Patients who acquire VAP have longer ICU stays, higher morbidity and mortality, and a greater number of infectious agents10,11. The risk factors for developing VAP are diverse, and the pathogenesis of intra-hospital infections is complex. Common VAP preventive measures such as early mobility, the daily interruption of sedation, and a readiness-to-extubate assessment may not be applicable because of associated injuries such as severe chest trauma, intra-abdominal bleeding, and other organ damage. Hence, VAP diagnosis can be difficult in a setting of multiple trauma, and significant variations in the diagnosis and management of VAP remain8.

The upper respiratory tract of the majority of mechanically-ventilated patient is colonized with potentially pathogenic microorganisms. This was first established in a study in 1969 that reported the presence of enteric gram-negative bacteria in the oropharynx of 75 percent of critically ill patients8. A proposed explanation is bacterial overgrowth of the upper gastrointestinal tract and retrograde movement. Aspiration of secretions containing these pathogens provides a means for infection of the sterile bronchial tree. Another study published in 2007 confirmed the presence of similar pathogenic microorganisms in the lower respiratory tract of intubated patients by comparing DNA samples from bacteria on the tongue and obtained from bronchoalveolar lavage (BAL)12.

Prevention of VAP:

The use of Non-invasive positive pressure ventilation NPPV has been shown to significantly lower the risk of VAP and has also demonstrated a mortality benefit in randomized studies conducted using patients with a variety of illnesses10, daily weaning trials and sedation holidays have been repeatedly described and validated as strategies that limit the time of mechanical ventilation13,14.

re-intubation is associated with a higher risk of VAP due to higher rates of aspiration15, It was previously thought that early tracheostomy might lead to better outcomes16.

Antimicrobial-coated endotracheal tubes (ETT) have been studied as a means to decrease bacterial colonization and prevent biofilm production with the ultimate hope of reducing VAP rates.

It is hypothesized that microorganisms reach the ETT either as a consequence of a contaminated oropharynx or reflux of gastric secretions29, selective digestive tract decontamination (SDD) and selective oropharyngeal decontamination (SoD) are measures in which antibiotic therapy is used to eradicate potentially pathogenic microorganisms in oral, gastric, and intestinal flora 17, 18.

Subglottic suctioning endotracheal tubes: It has been postulated that intermittently or continuously removing the secretions that pool above the ETT cuff may reduce the risk for aspiration and subsequent development of VAP. ETTs have therefore, been designed to accomplish this task through application of negative pressure to a separate port that opens above the ETT cuff19 Oral decontamination: Chlorhexidine is the oral antiseptic most rigorously studied with regards to VAP20, Iseganan and povidone iodine have also been investigated for oral decontamination. Iseganan is a topical antimicrobial with activity against grampositive and gram-negative bacteria, and yeast21 Elevation of the head of the bed is attempted to reduce aspiration of gastric content. The basis for this intervention comes from studies using radiolabelled enteral feeding solutions which have shown that aspiration of gastric contents occurs to a greater extent in supine patients than in patients in a semirecumbent position22,23 The goal of infection control is to prevent cross transmission of pathogens, which has been shown to play an important role in the development of nosocomial infections including VAP. An effective strategy should target infection control from several vantage points: education of the medical team, universal hand hygiene, use of personal protective equipment and a protocol for microbiological surveillance24

ELIGIBILITY:
Inclusion Criteria:

* - All patients with TBI who are on MV for >48 h after the initial evaluation.
* Patients are transferred either from the emergency room directly to the ICU, or they are transferred to the operating room first and are then admitted to the ICU after surgery.
* Patients intubated outside the hospital and who had no side effects are also included.

Exclusion Criteria:

* - Patients with documented gastric aspiration, recent antibiotic therapy, 2 days of hospitalization in the preceding 30 days, residence in a nursing home or extended care facility, home therapy, or an underlying malignancy are excluded.
* Patients who are transferred within the hospital if there was an accident or change in the ventilator system, or who have other known risk factors for developing pneumonia, are also excluded.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients are divided into three groups, as follows: patients who donot develop VAP, those who develop early onset VAP, and those who develop late-onset VAP with no age or sex predliction
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Risk factors and common preventive measures for ventilator associated pneumonia in patients with severe traumatic brain injury Risk factors and common preventive measures for ventilator associated pneumonia in patients with severe traumatic brain injury | all patients admitted to general or trauma ICU in assiut university hospital will be recorded from january 2018 to december 2018
  The patients are divided into three groups, as follows: patients who donot develop VAP, those who develop early onset VAP, and those who develop late-onset VAP
  • The primary objective of this study is to assess the incidence of VAP in patients with TBI and to identify risk factors for developing VAP in this specific patient population (types of co-injuries in patients with multiple trauma or characteristics on admission). The secondary objective is to assess the prevalence of pathogens responsible for early- and late-onset VAP in patients with TBI. The tertiary objective is to discuss the ability of preventive measures to reduce the incidence of VAP.